CLINICAL TRIAL: NCT01817530
Title: A Phase 2b Study to Evaluate the Safety and Efficacy of Elagolix in Premenopausal Women With Heavy Menstrual Bleeding Associated With Uterine Fibroids
Brief Title: Safety and Efficacy in Premenopausal Women With Heavy Menstrual Bleeding (HMB) Associated With Uterine Fibroids (UF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M12-813; 2013-000082-37 (EudraCT Number)
Record Dates: First submitted 2013-03-21; First posted 2013-03-25 (Estimated); Results first posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-06

CONDITIONS: Heavy Uterine Bleeding; Uterine Fibroids
Keywords: Uterine Fibroids; Leiomyomata; Elagolix; Menorrhagia; Elagolix sodium; Heavy Uterine Bleeding; ABT-620
MeSH Terms: conditions — Leiomyoma; Menorrhagia | interventions — elagolix; Estradiol; Norethindrone Acetate; estradiol, norethindrone drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1: Placebo (Placebo Comparator): Placebo for elagolix and placebo for E2/NETA twice daily (BID)
  Interventions: Other: Elagolix placebo; Drug: E2/NETA placebo
- Cohort 1: Elagolix 300 mg BID (Experimental): Elagolix 300 mg BID alone
  Interventions: Drug: Elagolix; Drug: E2/NETA placebo
- Cohort 1: Elagolix 300 mg BID plus LD E2/NETA QD (Experimental): Elagolix 300 mg BID plus low-dose (LD) E2/NETA once daily (QD)
  Interventions: Drug: Elagolix; Drug: 0.5 mg estradiol / 0.1 mg norethindrone acetate
- Cohort 1: Elagolix 300 mg BID plus SD E2/NETA QD (Experimental): Elagolix 300 mg BID plus standard-dose (SD) E2/NETA QD
  Interventions: Drug: Elagolix; Drug: 1 mg estradiol / 0.5 mg norethindrone acetate
- Cohort 2: Placebo (Placebo Comparator): Placebo for elagolix and E2/NETA QD
  Interventions: Other: Elagolix placebo; Drug: E2/NETA placebo
- Cohort 2: Elagolix 600 mg QD (Experimental): Elagolix 600 mg QD alone
  Interventions: Drug: Elagolix; Drug: E2/NETA placebo
- Cohort 2: Elagolix 600 mg QD plus LD E2/NETA QD (Experimental): Elagolix 600 mg QD plus LD E2/NETA QD
  Interventions: Drug: Elagolix; Drug: 0.5 mg estradiol / 0.1 mg norethindrone acetate
- Cohort 2: Elagolix 600 mg QD plus SD E2/NETA QD (Experimental): Elagolix 600 mg QD plus SD E2/NETA QD
  Interventions: Drug: Elagolix; Drug: 1 mg estradiol / 0.5 mg norethindrone acetate

INTERVENTIONS:
Other: Elagolix placebo — oral coated tablet
  Arms: Cohort 1: Placebo; Cohort 2: Placebo
Drug: Elagolix — oral coated tablet
  Other Names: ABT-620
  Arms: Cohort 1: Elagolix 300 mg BID; Cohort 1: Elagolix 300 mg BID plus LD E2/NETA QD; Cohort 1: Elagolix 300 mg BID plus SD E2/NETA QD; Cohort 2: Elagolix 600 mg QD; Cohort 2: Elagolix 600 mg QD plus LD E2/NETA QD; Cohort 2: Elagolix 600 mg QD plus SD E2/NETA QD
Drug: 0.5 mg estradiol / 0.1 mg norethindrone acetate — oral hard capsule
  Other Names: Activelle, Activella, low dose (LD) E2/NETA
  Arms: Cohort 1: Elagolix 300 mg BID plus LD E2/NETA QD; Cohort 2: Elagolix 600 mg QD plus LD E2/NETA QD
Drug: 1 mg estradiol / 0.5 mg norethindrone acetate — oral hard capsule
  Other Names: Activelle; Activella; standard dose (SD) E2/NETA
  Arms: Cohort 1: Elagolix 300 mg BID plus SD E2/NETA QD; Cohort 2: Elagolix 600 mg QD plus SD E2/NETA QD
Drug: E2/NETA placebo — oral hard capsule
  Arms: Cohort 1: Elagolix 300 mg BID; Cohort 1: Placebo; Cohort 2: Elagolix 600 mg QD; Cohort 2: Placebo

SUMMARY:
This is a Phase 2b randomized, double-blind, placebo-controlled study evaluating the safety and efficacy of elagolix alone and in combination with add-back therapy versus placebo on heavy menstrual bleeding in premenopausal women 18 to 51 years of age with uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* Subject is pre-menopausal female 18 to 51 years of age at Screening.
* Subject has diagnosis of uterine fibroids documented by a Pelvic Ultrasound.
* Subject has heavy uterine bleeding associated with uterine fibroids.

Exclusion Criteria:

* Subject has had a myomectomy, uterine artery embolization or high intensity focused ultrasound for fibroid destruction within 6 months prior to Screening or endometrial ablation within 5 years prior to Screening.
* Subject has a history of osteoporosis or other metabolic bone disease.
* Subject shows evidence of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric (including depression, schizophrenia, bipolar disorder), or neurologic diseases or any uncontrolled medical illness such as uncontrolled type 2 diabetes. Subject has any history of attempted suicide.
* Subject has a history of clinically significant condition(s) including but not limited to: * Symptomatic Endometriosis * Epilepsy or seizures * Type 1 diabetes * Chronic kidney disease * Any cancer (except treated basal cell carcinoma of the skin), including breast or ovarian cancer or subject has taken any systemic cancer chemotherapy

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 571 (Actual)
Dates: Start 2013-04-08 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Owens, MD, Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Carr BR, Stewart EA, Archer DF, Al-Hendy A, Bradley L, Watts NB, Diamond MP, Gao J, Owens CD, Chwalisz K, Duan WR, Soliman AM, Dufek MB, Simon JA. Elagolix Alone or With Add-Back Therapy in Women With Heavy Menstrual Bleeding and Uterine Leiomyomas: A Randomized Controlled Trial. Obstet Gynecol. 2018 Nov;132(5):1252-1264. doi: 10.1097/AOG.0000000000002933. PMID 30303923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 571 female participants were enrolled into the study across 86 sites (5 sites in the UK, 4 in Chile, 2 in Canada, 4 in Puerto Rico, and 71 in the US).
Pre-assignment Details: Four participants were randomized in error; they were not dosed and were excluded from all analyses including demographic summaries.
Groups:
- Cohort 1: Placebo: Placebo for elagolix twice daily (BID) and placebo for E2/NETA once daily (QD)
- Cohort 1: Elagolix 300 mg BID: Elagolix 300 mg BID and placebo for E2/NETA QD
- Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD: Elagolix 300 mg BID plus low-dose (LD) E2/NETA QD
- Cohort 2: Placebo: Placebo for elagolix QD and placebo for E2/NETA QD
- Cohort 2: Elagolix 600 mg QD: Elagolix 600 mg QD and placebo for E2/NETA QD
Period: Overall Study
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Started (randomized and treated) | 65 | 65 | 64 | 65 | 78 | 77 | 76 | 77
Completed | 50 | 52 | 53 | 52 | 67 | 58 | 53 | 53
Not Completed | 15 | 13 | 11 | 13 | 11 | 19 | 23 | 24
Not completed — Exclusionary Medication Received | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 3 | 2 | 5 | 0 | 10 | 5 | 8
Not completed — Subject Noncompliant | 3 | 1 | 0 | 4 | 0 | 1 | 1 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 0
Not completed — Surgery or Invasive Intervention | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Consent Withdrawn by Subject | 3 | 4 | 7 | 3 | 5 | 3 | 3 | 10
Not completed — Lost to Follow-up | 1 | 4 | 2 | 1 | 3 | 2 | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Placebo: Placebo for elagolix BID and placebo for E2/NETA QD
- Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD: Elagolix 300 mg BID plus LD E2/NETA QD
- Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD: Elagolix 300 mg BID plus SD E2/NETA QD
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD | Total
Number analyzed (Participants) | 65 | 65 | 64 | 65 | 78 | 77 | 76 | 77 | 567
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (6.14) | 42.0 (4.76) | 43.0 (5.02) | 43.8 (4.66) | 42.3 (4.78) | 42.1 (4.93) | 41.1 (5.74) | 42.2 (5.40) | 42.3 (5.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 65 | 64 | 65 | 78 | 77 | 76 | 77 | 567
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Menstrual Blood Loss (MBL) Volume of < 80 mL at the Final Month and a ≥ 50% Reduction in MBL Volume From Baseline to the Final Month
Description: The percentage of participants meeting a composite endpoint consisting of these 2 bleeding assessments: a MBL Volume of < 80 mL at the Final Month and a ≥50% Reduction in MBL Volume from Baseline to the Final Month (last 28 days of treatment). Baseline is defined as the last qualified menstrual cycle during the screening period.
Time Frame: Baseline, Final Month (last 28 days of treatment)
Population: Modified Intent-to-Treat (ITT): randomized participants who received at least 1 dose of randomized, double-blind study drug in this study. Excludes participants with < 28 days of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 64 | 62 | 61 | 62 | 76 | 71 | 73 | 76
percentage of participants | 26.56 | 91.94 | 85.25 | 79.03 | 31.58 | 90.14 | 72.6 | 81.58
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic — P value for test of difference between each elagolix dose group and placebo is from a logistic regression model including treatment as the main effect and baseline as a covariate; Odds Ratio (OR) = 32.51, 95% CI 2-sided [11.12 to 95.05]
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 16.66, 95% CI 2-sided [6.72 to 41.3]
Statistical Analysis 4: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 5: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 11.13, 95% CI 2-sided [4.79 to 25.84]
Statistical Analysis 6: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 7: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 19.62, 95% CI 2-sided [7.81 to 49.27]
Statistical Analysis 8: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 9: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 6.02, 95% CI 2-sided [2.95 to 12.3]
Statistical Analysis 10: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 11: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 10.34, 95% CI 2-sided [4.79 to 22.34]
Statistical Analysis 12: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test

2. Secondary Outcome: Percentage of Participants With a MBL Volume < 80 mL and a ≥ 50% Reduction in MBL Volume From Baseline During the Last 56 to 29 Days of Treatment
Description: The percentage of participants meeting a composite endpoint consisting of these 2 bleeding assessments: a MBL volume < 80 mL and a ≥ 50% reduction in MBL volume from baseline during the last 56 to 29 days of last treatment. Baseline is defined as the last qualified menstrual cycle during the screening period.
Time Frame: Baseline, second last 28 days of treatment (last 56 to 29 days of treatment)
Population: Modified ITT: randomized participants who received at least 1 dose of randomized, double-blind study drug in this study. Excludes participants with < 56 days of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 62 | 58 | 59 | 60 | 76 | 68 | 64 | 70
percentage of participants | 11.29 | 94.83 | 88.14 | 85.00 | 18.42 | 85.29 | 67.19 | 77.14
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 156.17, 95% CI 2-sided [38.04 to 641.22]
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 66.07, 95% CI 2-sided [21.1 to 206.88]
Statistical Analysis 4: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 5: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 52.15, 95% CI 2-sided [17.42 to 156.09]
Statistical Analysis 6: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 7: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 25.45, 95% CI 2-sided [10.45 to 61.96]
Statistical Analysis 8: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 9: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 9.65, 95% CI 2-sided [4.38 to 21.25]
Statistical Analysis 10: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 11: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 16.17, 95% CI 2-sided [7.13 to 36.67]
Statistical Analysis 12: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test

3. Secondary Outcome: Percentage of Participants With a MBL Volume < 80 mL and a ≥ 50% Reduction in MBL Volume From Baseline During the Last 84 to 57 Days of Treatment
Description: The percentage of participants meeting a composite endpoint consisting of these 2 bleeding assessments: a MBL volume < 80 mL and a ≥ 50% reduction in MBL volume from baseline during the last 84 to 57 days of last treatment. Baseline is defined as the last qualified menstrual cycle during the screening period.
Time Frame: Baseline, third last 28 days of treatment (last 84 to 57 days of treatment)
Population: Modified ITT: randomized participants who received at least 1 dose of randomized, double-blind study drug in this study. Excludes participants with < 84 days of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 61 | 56 | 57 | 58 | 74 | 66 | 62 | 65
percentage of participants | 19.67 | 96.43 | 89.47 | 79.31 | 21.62 | 86.36 | 74.19 | 72.31
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 123.14, 95% CI 2-sided [25.93 to 584.85]
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 40.56, 95% CI 2-sided [13.59 to 121.03]
Statistical Analysis 4: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 5: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 19.01, 95% CI 2-sided [7.44 to 48.58]
Statistical Analysis 6: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 7: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 22.77, 95% CI 2-sided [9.29 to 55.77]
Statistical Analysis 8: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 9: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 10.89, 95% CI 2-sided [4.88 to 24.27]
Statistical Analysis 10: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 11: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 9.72, 95% CI 2-sided [4.46 to 21.22]
Statistical Analysis 12: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test

4. Secondary Outcome: Percentage of Participants Who Achieved an MBL Volume of < 80 mL at the Final Month
Description: Percentage of participants who achieved an MBL volume of < 80 mL at the Final Month (last 28 days of treatment). Baseline is defined as the last qualified menstrual cycle during the screening period.
Time Frame: Final Month (last 28 days of treatment)
Population: Modified ITT: randomized participants who received at least 1 dose of randomized, double-blind study drug in this study. Excludes participants with < 28 days of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 64 | 62 | 61 | 62 | 76 | 71 | 73 | 76
percentage of participants | 32.81 | 91.94 | 88.52 | 79.03 | 36.84 | 91.55 | 72.6 | 85.53
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic — P value for test of difference between each elagolix dose group and placebo is from a logistic regression model including treatment as the main effect and baseline value as a covariate; Odds Ratio (OR) = 24.73, 95% CI 2-sided [8.57 to 71.32]
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 17.21, 95% CI 2-sided [6.57 to 45.05]
Statistical Analysis 4: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 5: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 8.69, 95% CI 2-sided [3.79 to 19.92]
Statistical Analysis 6: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 7: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 18.67, 95% CI 2-sided [7.11 to 49.02]
Statistical Analysis 8: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 9: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 4.94, 95% CI 2-sided [2.43 to 10.04]
Statistical Analysis 10: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 11: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic; P value is from a logistic regression model including treatment as the main effect and baseline value as a covariate; Odds Ratio (OR) = 11.76, 95% CI 2-sided [5.17 to 26.79]
Statistical Analysis 12: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test

5. Secondary Outcome: Percentage of Participants With a ≥ 50% Reduction in MBL Volume From Baseline to the Final Month
Description: Percentage of participants with a >= 50% reduction from baseline in MBL to the Final Month (last 28 days of treatment). Baseline is defined as the last qualified menstrual cycle during the screening period.
Time Frame: Baseline, Final Month (last 28 days of treatment)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 64 | 62 | 61 | 62 | 76 | 71 | 73 | 76
percentage of participants | 31.25 | 93.55 | 86.89 | 82.26 | 35.53 | 90.14 | 79.45 | 85.53
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 31.48, 95% CI 2-sided [10.02 to 98.83]
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 14.39, 95% CI 2-sided [5.77 to 35.91]
Statistical Analysis 4: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 5: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 9.82, 95% CI 2-sided [4.23 to 22.8]
Statistical Analysis 6: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 7: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 16.58, 95% CI 2-sided [6.66 to 41.26]
Statistical Analysis 8: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 9: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 7.02, 95% CI 2-sided [3.36 to 14.68]
Statistical Analysis 10: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test
Statistical Analysis 11: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 10.73, 95% CI 2-sided [4.85 to 23.76]
Statistical Analysis 12: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Chi-squared — P value for test of difference between each elagolix dose group and placebo is from a chi-square test

6. Secondary Outcome: Percentage of Participants Who Achieved Amenorrhea During the Last 56 Days of Treatment
Description: Amenorrhea is defined as having 0 days of bleeding or spotting based on observed validated and nonvalidated alkaline hematin data and having 0 days of bleeding or spotting, based on imputed electronic diary data during the last 56 days of treatment. Participants needed to have at least 66 days on treatment.
Time Frame: Last 56 days of treatment (after 10 days from first dose date)
Population: Modified ITT: randomized participants who received at least 1 dose of randomized, double-blind study drug in this study. Excludes participants with < 66 days of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 61 | 57 | 57 | 60 | 75 | 67 | 63 | 66
percentage of participants | 1.6 | 56.1 | 33.3 | 28.3 | 1.3 | 50.7 | 17.5 | 22.7
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 5: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 6: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Fisher Exact

7. Secondary Outcome: Percentage of Participants Who Achieved Suppression of Bleeding During the Last 56 Days of Treatment
Description: Suppression of bleeding is defined as having 0 days of bleeding based on observed validated and nonvalidated alkaline hematin data and having 0 days of bleeding (spotting is allowed) based on imputed electronic diary data during the last 56 days of treatment.
Time Frame: Last 56 days of treatment (after 10 days from first dose date)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 61 | 57 | 57 | 60 | 75 | 67 | 63 | 66
percentage of participants | 1.6 | 75.4 | 52.6 | 43.3 | 2.7 | 67.2 | 31.7 | 34.8
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 5: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 6: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, Fisher Exact

8. Secondary Outcome: Mean Change in the Number of Bleeding Days From Baseline to Month 6
Description: The number of days with any bleeding including spotting was calculated using data collected on daily bleeding diary. Baseline is defined as the last 28 days prior to the first dose day of study drug.
Time Frame: Baseline, Month 6
Population: Modified ITT: randomized participants who received at least 1 dose of randomized, double-blind study drug in this study. Participants with an assessment at baseline and Month 6.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 37 | 11 | 26 | 30 | 47 | 15 | 26 | 28
days | -1.2 (0.63) | -4.9 (1.15) | -2.7 (0.75) | -1.1 (0.69) | -1.4 (0.49) | -3.3 (0.87) | -1.3 (0.66) | -1.8 (0.64)
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p = 0.007, ANCOVA — P value for test of difference between each elagolix dose group and placebo at each postbaseline time point is from an ANCOVA model with treatment as the main effect and baseline value as a covariate; difference in LS mean change = -3.7, 95% CI 2-sided [-6.28 to -1.03], Standard Error of Mean 1.32
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p = 0.132, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS mean change = -1.5, 95% CI 2-sided [-3.44 to 0.46], Standard Error of Mean 0.98
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p = 0.876, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS mean change = 0.1, 95% CI 2-sided [-1.71 to 2.00], Standard Error of Mean 0.94
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p = 0.055, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS mean change = -1.9, 95% CI 2-sided [-3.92 to 0.04], Standard Error of Mean 1.00
Statistical Analysis 5: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p = 0.898, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS mean change = 0.1, 95% CI 2-sided [-1.52 to 1.74], Standard Error of Mean 0.82
Statistical Analysis 6: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p = 0.59, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS mean change = -0.4, 95% CI 2-sided [-2.05 to 1.17], Standard Error of Mean 0.81

9. Secondary Outcome: Mean Change in the Number of Heavy Bleeding Days From Baseline to Month 6
Description: The number of days with heavy bleeding (either heavy or very heavy/gushing bleeding) was calculated using data collected on daily bleeding diary. Baseline is defined as the last 28 days prior to the first dose day of study drug.
Time Frame: Baseline, Month 6
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 37 | 11 | 26 | 30 | 47 | 15 | 26 | 28
days | -1.0 (0.15) | -2.0 (0.27) | -1.9 (0.18) | -1.7 (0.16) | -0.7 (0.14) | -1.2 (0.25) | -1.4 (0.19) | -1.8 (0.18)
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p = 0.001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS mean change = -1.00, 95% CI 2-sided [-1.64 to -0.42], Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS mean change = -1.00, 95% CI 2-sided [-1.42 to -0.48], Standard Error of Mean 0.23
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p = 0.002, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS mean change = -0.7, 95% CI 2-sided [-1.12 to -0.25], Standard Error of Mean 0.22
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p = 0.118, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS mean change = -0.5, 95% CI 2-sided [-1.04 to 0.12], Standard Error of Mean 0.29
Statistical Analysis 5: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p = 0.004, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS mean change = -0.7, 95% CI 2-sided [-1.16 to -0.22], Standard Error of Mean 0.24
Statistical Analysis 6: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS mean change = -1.00, 95% CI 2-sided [-1.51 to -0.59], Standard Error of Mean 0.23

10. Secondary Outcome: Change in Bleeding Severity Scores From Baseline at the Final Month
Description: The average bleeding score was calculated for each 28-day interval starting on Day 29 using data collected on daily bleeding diary using the Mansfield-Voda-Jorgenson (MVJ) Menstrual Bleeding Scale (1=spotting, 2 = very light bleeding, 3 = light bleeding, 4 = moderate bleeding, 5 = heavy bleeding, 6 = very heavy/gushing bleeding). Baseline is defined as the last 28 days prior to the first day of study drug.
Time Frame: Baseline, Final Month (last 28 days of treatment)
Population: Modified ITT: randomized participants who received at least 1 dose of randomized, double-blind study drug in this study. Participants with an assessment at baseline and final month.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 51 | 19 | 33 | 37 | 61 | 24 | 48 | 42
units on a scale | -0.3 (0.08) | -0.7 (0.14) | -0.4 (0.10) | -0.1 (0.10) | -0.2 (0.08) | -0.4 (0.14) | -0.3 (0.10) | -0.1 (0.10)
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p = 0.004, ANCOVA — P value for test of difference between each elagolix dose group and placebo at each post-baseline time point is from an ANCOVA model with treatment as the main effect and baseline as a covariate; difference in LS mean change = -0.5, 95% CI 2-sided [-0.79 to -0.15], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p = 0.314, ANCOVA — [p-value comment as in outcome 10, analysis 1]; difference in LS mean change = -0.1, 95% CI 2-sided [-0.4 to 0.13], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p = 0.307, ANCOVA — [p-value comment as in outcome 10, analysis 1]; difference in LS mean change = 0.1, 95% CI 2-sided [-0.12 to 0.39], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p = 0.106, ANCOVA — [p-value comment as in outcome 10, analysis 1]; difference in LS mean change = -0.3, 95% CI 2-sided [-0.58 to 0.06], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p = 0.424, ANCOVA — [p-value comment as in outcome 10, analysis 1]; difference in LS mean change = -0.1, 95% CI 2-sided [-0.36 to 0.15], Standard Error of Mean 0.13
Statistical Analysis 6: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p = 0.528, ANCOVA — [p-value comment as in outcome 10, analysis 1]; difference in LS mean change = 0.1, 95% CI 2-sided [-0.18 to 0.35], Standard Error of Mean 0.13

11. Secondary Outcome: Mean Change in Hemoglobin Concentration From Baseline to Final Visit
Description: Baseline is defined as the last measurement prior to the first dose of study drug.
Time Frame: Baseline, Final Visit during treatment period (Month 6 or early termination)
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 64 | 61 | 59 | 61 | 76 | 71 | 72 | 74
g/dL | 0.6 (0.17) | 1.9 (0.17) | 1.9 (0.17) | 1.4 (0.17) | 0.3 (0.15) | 1.4 (0.16) | 1.1 (0.16) | 1.2 (0.16)
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS means = 1.3, 95% CI 2-sided [0.80 to 1.74], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS means = 1.3, 95% CI 2-sided [0.78 to 1.72], Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS means = 0.8, 95% CI 2-sided [0.33 to 1.27], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS means = 1.1, 95% CI 2-sided [0.65 to 1.52], Standard Error of Mean 0.22
Statistical Analysis 5: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS means = 0.7, 95% CI 2-sided [0.29 to 1.16], Standard Error of Mean 0.22
Statistical Analysis 6: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; difference in LS means = 0.8, 95% CI 2-sided [0.4 to 1.26], Standard Error of Mean 0.22

12. Secondary Outcome: Mean Percentage Change From Baseline in Total Fibroid Volume at Month 3, Month 6, and Final Visit
Description: Volume of the total fibroid volume (3 largest fibroids), as measured by transvaginal ultrasound, or transabdominal ultrasound.
Time Frame: Baseline, Month 3, Month 6, and Final Visit during treatment period (Month 6 or early termination)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 65 | 65 | 64 | 65 | 78 | 77 | 76 | 77
percentage change
  Month 3: number analyzed (Participants) | 53 | 49 | 52 | 47 | 64 | 57 | 53 | 58
  Month 3 | 1.7 (33.61) | -41.9 (24.87) | -24.6 (27.58) | -9.8 (40.31) | 5.4 (27.18) | -34.4 (25.56) | -17.5 (27.76) | -4.6 (39.97)
  Month 6: number analyzed (Participants) | 45 | 44 | 48 | 42 | 55 | 50 | 44 | 46
  Month 6 | 8.3 (50.97) | -40.2 (27.6) | -23.3 (30.34) | -8.8 (47.81) | -1.8 (30.1) | -34.2 (31.14) | -17.8 (30.49) | -1.1 (46.66)
  Final Visit: number analyzed (Participants) | 53 | 53 | 54 | 51 | 66 | 59 | 55 | 60
  Final Visit | 4.6 (48.59) | -39.6 (28.66) | -24.0 (29.93) | -12.9 (46.2) | 0.1 (28.82) | -36.4 (30.07) | -16.6 (32.65) | -1.6 (42.75)
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Month 3; Test type: Superiority; p < 0.001, Kruskal-Wallis — P value for test of difference between each elagolix dose group and placebo is from Kruskal-Wallis analysis with treatment as the main effect
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Month 3; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Month 3; Test type: Superiority; p = 0.018, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Month 3; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 5: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Month 3; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 6: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Month 3; Test type: Superiority; p = 0.021, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 7: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Month 6; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 8: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Month 6; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 9: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Month 6; Test type: Superiority; p = 0.032, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 10: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Month 6; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 11: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Month 6; Test type: Superiority; p = 0.007, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 12: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Month 6; Test type: Superiority; p = 0.495, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 13: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Final Visit; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 14: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Final Visit; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 15: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Final Visit; Test type: Superiority; p = 0.015, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 16: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Final Visit; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 17: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Final Visit; Test type: Superiority; p = 0.002, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 18: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Final Visit; Test type: Superiority; p = 0.329, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]

13. Secondary Outcome: Mean Percentage Change From Baseline in Primary Fibroid Volume at Month 3, Month 6, and Final Visit
Description: Volume of the largest fibroid (primary fibroid), as measured by transvaginal ultrasound, or transabdominal ultrasound.
Time Frame: Baseline, Month 3, Month 6, and Final Visit during treatment period (Month 6 or early termination)
Population: Modified ITT: randomized participants who received at least 1 dose of randomized, double-blind study drug in this study. Participants with an assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 65 | 65 | 64 | 65 | 78 | 77 | 76 | 77
percentage change
  Month 3: number analyzed (Participants) | 53 | 49 | 52 | 47 | 64 | 57 | 53 | 58
  Month 3 | 6.9 (35.31) | -35.5 (26.32) | -20.3 (33.54) | -3.7 (39.13) | 6.7 (27.66) | -33.6 (23.74) | -17.2 (27.39) | -1.9 (39.22)
  Month 6: number analyzed (Participants) | 45 | 44 | 48 | 42 | 55 | 50 | 44 | 46
  Month 6 | 13.2 (48.65) | -36.1 (30.59) | -19.6 (32.1) | 0.0 (47.07) | 1.4 (30.03) | -33.5 (31.89) | -12.2 (40.59) | -0.7 (42.98)
  Final Visit: number analyzed (Participants) | 53 | 53 | 54 | 51 | 66 | 59 | 55 | 60
  Final Visit | 9.0 (46.63) | -35.6 (30.81) | 20.0 (31.73) | -2.7 (46.63) | 3.0 (28.7) | -34.8 (30.36) | -12.8 (39.65) | 0.0 (40.17)
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Month 3; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Month 3; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Month 3; Test type: Superiority; p = 0.036, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Month 3; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 5: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Month 3; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 6: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Test type: Superiority; p = 0.040, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 7: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Month 6; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 8: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 9: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Month 6; Test type: Superiority; p = 0.098, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 10: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Month 6; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 11: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Month 6; Test type: Superiority; p = 0.014, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 12: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Month 6; Test type: Superiority; p = 0.409, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 13: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Final Visit; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 14: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Final Visit; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 15: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Final Visit; Test type: Superiority; p = 0.094, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 16: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Final Visit; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 17: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Final Visit; Test type: Superiority; p = 0.002, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 18: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Final Visit; Test type: Superiority; p = 0.393, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]

14. Secondary Outcome: Mean Percentage Change From Baseline in Uterine Volume at Month 3, Month 6, and Final Visit
Description: Uterine volume, as measured by transvaginal ultrasound or transabdominal ultrasound.
Time Frame: Baseline, Month 3, Month 6, and Final Visit during treatment period (Month 6 or early termination)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 65 | 65 | 64 | 65 | 78 | 77 | 76 | 77
percentage change
  Month 3: number analyzed (Participants) | 58 | 52 | 56 | 54 | 72 | 63 | 57 | 63
  Month 3 | 7.3 (25.12) | -30.9 (28.87) | -19.4 (22.48) | -7.3 (20.7) | 8.4 (24.26) | -24.7 (21.98) | -15.7 (21.84) | -6.1 (18.81)
  Month 6: number analyzed (Participants) | 51 | 47 | 50 | 47 | 61 | 56 | 49 | 50
  Month 6 | 17.5 (40.25) | -35.6 (25.74) | -21.9 (27.64) | -13.2 (23.86) | 10.7 (20.73) | -26.00 (29.51) | -13.5 (25.09) | -9.0 (22.12)
  Final Visit: number analyzed (Participants) | 58 | 56 | 56 | 56 | 72 | 65 | 58 | 64
  Final Visit | 15.9 (38.06) | -31.5 (31.44) | -22.0 (28.52) | -11.8 (22.56) | 11.6 (25.38) | -26.6 (28.26) | -11.5 (25.33) | -6.7 (21.8)
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Month 3; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Month 3; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Month 3; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Month 3; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 5: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Month 3; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 6: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Month 6; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 7: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Month 6; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 8: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Month 6; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 9: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Month 6; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 10: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Month 6; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 11: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Month 6; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 12: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Final Visit; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 13: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Final Visit; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 14: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Final Visit; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 15: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Final Visit; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 16: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Final Visit; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 17: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Final Visit; Test type: Superiority; p < 0.001, Kruskal-Wallis — [p-value comment as in outcome 12, analysis 1]

15. Secondary Outcome: Percentage of Participants With ≥ 25% Reduction From Baseline in Total Fibroid Volume at Month 3, Month 6, and Final Visit
Description: Total fibroid volume (3 largest fibroids) was measured by transvaginal ultrasound, or transabdominal ultrasound.
Time Frame: Baseline, Month 3, Month 6, and Final Visit during treatment period (Month 6 or early termination)
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 65 | 65 | 64 | 65 | 78 | 77 | 76 | 77
percentage of participants
  Month 3: number analyzed (Participants) | 53 | 49 | 52 | 47 | 64 | 57 | 53 | 58
  Month 3 | 13.2 | 79.6 | 50.0 | 31.9 | 9.4 | 66.7 | 34.0 | 22.4
  Month 6: number analyzed (Participants) | 45 | 44 | 48 | 42 | 55 | 50 | 44 | 46
  Month 6 | 24.4 | 75.0 | 54.2 | 40.5 | 18.2 | 62.0 | 40.9 | 34.8
  Final Visit: number analyzed (Participants) | 53 | 53 | 54 | 51 | 66 | 59 | 55 | 60
  Final Visit | 24.5 | 73.6 | 57.4 | 41.2 | 16.7 | 64.4 | 40.0 | 30.0
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Month 3; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Month 3; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Month 3; Test type: Superiority; p = 0.020, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Month 3; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Month 3; Test type: Superiority; p = 0.002, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Month 3; Test type: Superiority; p = 0.061, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Month 6; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Month 6; Test type: Superiority; p = 0.004, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Month 6; Test type: Superiority; p = 0.085, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Month 6; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 11: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Month 6; Test type: Superiority; p = 0.012, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 12: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Month 6; Test type: Superiority; p = 0.049, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 13: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Final Visit; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 14: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Final Visit; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 15: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Final Visit; Test type: Superiority; p = 0.056, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 16: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Final Visit; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 17: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Final Visit; Test type: Superiority; p = 0.005, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 18: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Final Visit; Test type: Superiority; p = 0.088, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]

16. Secondary Outcome: Percentage of Participants With ≥ 25% Reduction From Baseline in Primary Fibroid Volume at Month 3, Month 6, and Final Visit
Description: Volume of the largest fibroid (primary fibroid) was measured by transvaginal ultrasound or transabdominal ultrasound.
Time Frame: Baseline, Month 3, Month 6, and Final Visit during treatment period (Month 6 or early termination)
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 65 | 65 | 64 | 65 | 78 | 77 | 76 | 77
percentage of participants
  Month 3: number analyzed (Participants) | 53 | 49 | 52 | 47 | 64 | 57 | 53 | 58
  Month 3 | 13.2 | 67.3 | 46.2 | 23.4 | 10.9 | 63.2 | 37.7 | 22.4
  Month 6: number analyzed (Participants) | 45 | 44 | 48 | 42 | 55 | 50 | 44 | 46
  Month 6 | 24.4 | 70.5 | 47.9 | 26.2 | 14.5 | 64.0 | 38.6 | 34.8
  Final Visit: number analyzed (Participants) | 53 | 53 | 54 | 51 | 66 | 59 | 55 | 60
  Final Visit | 24.5 | 69.8 | 50.0 | 27.5 | 13.6 | 66.1 | 40.0 | 30.0
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Month 3; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Month 3; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Month 3; Test type: Superiority; p = 0.188, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Month 3; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Month 3; Test type: Superiority; p = 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Month 3; Test type: Superiority; p = 0.104, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Month 6; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Month 6; Test type: Superiority; p = 0.021, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Month 6; Test type: Superiority; p = 0.859, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Month 6; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 11: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Month 6; Test type: Superiority; p = 0.006, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 12: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Month 6; Test type: Superiority; p = 0.015, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 13: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Final Visit; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 14: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Final Visit; Test type: Superiority; p = 0.007, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 15: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Final Visit; Test type: Superiority; p = 0.722, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 16: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Final Visit; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 17: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Final Visit; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 18: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Final Visit; Test type: Superiority; p = 0.032, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]

17. Secondary Outcome: Percentage of Participants With ≥ 25% Reduction From Baseline in Uterine Volume at Month 3, Month 6, and Final Visit
Description: Uterine volume was measured by transvaginal ultrasound or transabdominal ultrasound.
Time Frame: Baseline, Month 3, Month 6, and Final Visit during treatment period (Month 6 or early termination)
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 65 | 65 | 64 | 65 | 78 | 77 | 76 | 77
percentage of participants
  Month 3: number analyzed (Participants) | 58 | 52 | 56 | 54 | 72 | 63 | 57 | 63
  Month 3 | 5.2 | 73.1 | 42.9 | 18.5 | 1.4 | 57.1 | 36.8 | 17.5
  Month 6: number analyzed (Participants) | 51 | 47 | 50 | 47 | 61 | 56 | 49 | 50
  Month 6 | 2.0 | 78.7 | 58.0 | 31.9 | 1.6 | 62.5 | 32.7 | 26.0
  Final Visit: number analyzed (Participants) | 58 | 56 | 56 | 56 | 72 | 65 | 58 | 64
  Final Visit | 3.4 | 73.2 | 58.9 | 26.8 | 1.4 | 63.1 | 29.3 | 23.4
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Month 3; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Month 3; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Month 3; Test type: Superiority; p = 0.041, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Month 3; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Month 3; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Month 3; Test type: Superiority; p = 0.008, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Month 6; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Month 6; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Month 6; Test type: Superiority; p = 0.003, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Month 6; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 11: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Month 6; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 12: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Month 6; Test type: Superiority; p = 0.003, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 13: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Final Visit; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 14: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Final Visit; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 15: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Final Visit; Test type: Superiority; p = 0.004, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 16: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Final Visit; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 17: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Final Visit; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 18: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Final Visit; Test type: Superiority; p = 0.002, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]

18. Secondary Outcome: Change From Baseline to Each Month in Non-Bleeding Uterine Fibroids Symptom (NBUFSQ) Questionnaire
Description: The NBUFSQ (8 items) is a brief patient-reported daily diary that assesses non-bleeding symptoms experienced by women with uterine fibroids. It includes 6 items, asking women to rate their symptoms (abdominal/pelvic pain, pressure, and cramping, back pain, bloating, and urinary problems) in the past 24 hours using an 11-point numeric response scale that ranges from 0 (i.e., no symptom) to 10 (i.e., worst possible symptom) and 2 items to address urinary frequency during the daytime and at night. Data presented in the sum of scores to the 6 symptom questions, ranging from 0 (no symptoms) to 60 (worst possible symptoms). Baseline is defined as the last 28 days prior to the first day of study drug. Final Month is defined as the last 28 days prior to and including the last dose date of study drug.
Time Frame: Baseline, Days 1-28, Days 29-56, Days 57-84, Days 85-112, Days 113-140, Days 141-168, Final Month of treatment, Post-treatment (PT) Days 1-28, PT Days 29-56, PT Days 57-84, PT Days 85-112, PT Days 113-140, PT Days 141-168
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 65 | 65 | 64 | 65 | 78 | 77 | 76 | 77
units on a scale
  Days 1-28: number analyzed (Participants) | 37 | 36 | 36 | 34 | 71 | 74 | 71 | 67
  Days 1-28 | -3.3 (10.11) | -3.4 (8.21) | -3.1 (7.88) | -1.4 (6.42) | 0.4 (4.71) | -2.7 (7.27) | -2.1 (4.44) | 0.0 (6.26)
  Days 29-56: number analyzed (Participants) | 35 | 34 | 34 | 28 | 68 | 65 | 63 | 63
  Days 29-56 | -4.5 (13.12) | -5.8 (8.78) | -4.4 (6.59) | -2.9 (9.44) | -0.3 (7.13) | -4.2 (7.72) | -2.2 (5.54) | -2.3 (9.31)
  Days 57-84: number analyzed (Participants) | 34 | 31 | 34 | 28 | 61 | 63 | 56 | 54
  Days 57-84 | -5.6 (10.94) | -7.2 (11.04) | -4.1 (8.4) | -3.2 (11.26) | 0.1 (7.34) | -4.5 (8.55) | -2.2 (6.22) | -3.8 (8.92)
  Days 85-112: number analyzed (Participants) | 31 | 31 | 31 | 28 | 55 | 62 | 55 | 53
  Days 85-112 | -7.0 (10.74) | -7.8 (11.75) | -5.2 (9.05) | -3.7 (10.76) | -0.2 (7.47) | -5.1 (9.40) | -3.6 (7.35) | -4.1 (8.96)
  Days 113-140: number analyzed (Participants) | 28 | 29 | 32 | 28 | 56 | 57 | 48 | 47
  Days 113-140 | -4.1 (13.16) | -7.6 (12.03) | -5.3 (9.43) | -3.4 (12.1) | 0.1 (11.92) | -5.5 (8.44) | -4.0 (8.13) | -5.3 (8.99)
  Days 141-168: number analyzed (Participants) | 26 | 29 | 30 | 27 | 53 | 51 | 47 | 45
  Days 141-168 | -6.8 (14.28) | -8.0 (12.65) | -5.1 (9.94) | -3.3 (13.01) | -0.4 (10.46) | -5.9 (9.45) | -4.4 (8.21) | -4.8 (9.3)
  Final Month: number analyzed (Participants) | 37 | 34 | 33 | 31 | 66 | 70 | 65 | 61
  Final Month | -5.3 (13.19) | -6.7 (11.94) | -4.1 (10.15) | -3.5 (12.59) | -0.8 (11.34) | -4.0 (9.40) | -3.3 (8.09) | -2.3 (10.56)
  PT Days 1-28: number analyzed (Participants) | 29 | 30 | 28 | 27 | 61 | 63 | 59 | 57
  PT Days 1-28 | -5.6 (13.39) | -5.2 (12.13) | -3.8 (10.37) | -3.0 (10.69) | -0.8 (12.46) | -3.8 (10.53) | -2.0 (8.23) | -2.3 (7.82)
  PT Days 29-56: number analyzed (Participants) | 28 | 29 | 30 | 26 | 59 | 58 | 53 | 53
  PT Days 29-56 | -5.7 (15.83) | -4.1 (13.1) | -1.0 (11.57) | 0.0 (9.89) | -0.2 (12.49) | -2.8 (11.85) | -2.7 (7.58) | -2.5 (8.54)
  PT Days 57-84: number analyzed (Participants) | 26 | 27 | 27 | 24 | 58 | 55 | 49 | 47
  PT Days 57-84 | -5.4 (17.08) | -4.0 (14.11) | -2.1 (10.91) | -1.1 (10.50) | -0.5 (13.08) | -2.0 (9.79) | -1.6 (8.35) | -3.9 (6.87)
  PT Days 85-112: number analyzed (Participants) | 12 | 10 | 10 | 11 | 23 | 26 | 23 | 19
  PT Days 85-112 | -4.4 (17.82) | -6.4 (12.99) | -4.8 (10.33) | 0.7 (6.59) | -2.7 (7.15) | -2.4 (14.37) | -3.0 (7.48) | -5.0 (5.12)
  PT Days 113-140: number analyzed (Participants) | 4 | 2 | 1 | 3 | 4 | 4 | 4 | 3
  PT Days 113-140 | 3.4 (27.8) | -3.1 (2.15) | 1.3 (NA) — only 1 participant analyzed | 1.4 (1.75) | -6.2 (1.51) | -17.3 (26.2) | -5.6 (6.45) | -7.0 (7.12)
  PT Days 141-168: number analyzed (Participants) | 3 | 2 | 1 | 1 | 1 | 1 | 4 | 3
  PT Days 141-168 | 7.5 (27.75) | -8.0 (1.42) | 4.1 (NA) — only 1 participant analyzed | -3.3 (NA) — only 1 participant analyzed | -10.5 (NA) — only 1 participant analyzed | -3.1 (NA) — only 1 participant analyzed | -3.3 (6.42) | -6.4 (5.94)
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID; Final Month; Test type: Superiority; p = 0.556, ANCOVA — P value for test of difference between each elagolix dose group and placebo at each post-baseline time point is from ANCOVA model with treatment as the main effect and baseline as covariate; difference in LS means = -1.5, 95% CI 2-sided [-6.65 to 3.59], Standard Error of Mean 2.58
Statistical Analysis 2: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD; Final Month; Test type: Superiority; p = 0.672, ANCOVA — [p-value comment as in outcome 18, analysis 1]; difference in LS means = -1.1, 95% CI 2-sided [-6.33 to 4.09], Standard Error of Mean 2.63
Statistical Analysis 3: Comparison: Cohort 1: Placebo vs Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD; Final Month; Test type: Superiority; p = 0.274, ANCOVA — [p-value comment as in outcome 18, analysis 1]; difference in LS means = 3.0, 95% CI 2-sided [-2.39 to 8.36], Standard Error of Mean 2.71
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD; Final Month; Test type: Superiority; p = 0.223, ANCOVA — [p-value comment as in outcome 18, analysis 1]; difference in LS means = -2.0, 95% CI 2-sided [-5.26 to 1.23], Standard Error of Mean 1.65
Statistical Analysis 5: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD; Final Month; Test type: Superiority; p = 0.215, ANCOVA — [p-value comment as in outcome 18, analysis 1]; difference in LS means = -2.1, 95% CI 2-sided [-5.38 to 1.22], Standard Error of Mean 1.68
Statistical Analysis 6: Comparison: Cohort 2: Placebo vs Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD; Final Month; Test type: Superiority; p = 0.392, ANCOVA — [p-value comment as in outcome 18, analysis 1]; difference in LS means = -1.4, 95% CI 2-sided [-4.75 to 1.87], Standard Error of Mean 1.68

19. Secondary Outcome: Percentage of Participants Who Successfully Avoided Surgical or Invasive Procedures for Uterine Fibroids
Description: The percentage of participants who successfully avoided surgical or invasive procedures for Uterine Fibroids was assessed.
Time Frame: Month 6
Population: This endpoint was not completed due to lack of data collection.
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of study drug administration through Final Visit (Month 6 or early termination) plus 30 days
Arm/Group | Cohort 1: Placebo | Cohort 1: Elagolix 300 mg BID | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD | Cohort 2: Placebo | Cohort 2: Elagolix 600 mg QD | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65 | 0/64 | 0/65 | 0/78 | 0/77 | 0/76 | 0/77
Serious Adverse Events (participants affected / at risk) | 6/65 | 3/65 | 3/64 | 1/65 | 1/78 | 5/77 | 3/76 | 4/77
Other Adverse Events (participants affected / at risk) | 33/65 | 45/65 | 37/64 | 44/65 | 42/78 | 59/77 | 43/76 | 51/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Placebo (N=65) | Cohort 1: Elagolix 300 mg BID (N=65) | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD (N=64) | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD (N=65) | Cohort 2: Placebo (N=78) | Cohort 2: Elagolix 600 mg QD (N=77) | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD (N=76) | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD (N=77)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VARICELLA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRINOMA MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CYSTOCELE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MENORRHAGIA (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Placebo (N=65) | Cohort 1: Elagolix 300 mg BID (N=65) | Cohort 1: Elagolix 300 mg BID Plus LD E2/NETA QD (N=64) | Cohort 1: Elagolix 300 mg BID Plus SD E2/NETA QD (N=65) | Cohort 2: Placebo (N=78) | Cohort 2: Elagolix 600 mg QD (N=77) | Cohort 2: Elagolix 600 mg QD Plus LD E2/NETA QD (N=76) | Cohort 2: Elagolix 600 mg QD Plus SD E2/NETA QD (N=77)
ANAEMIA (Blood and lymphatic system disorders) | 6 (6) | 1 (1) | 2 (2) | 2 (2) | 6 (6) | 3 (3) | 6 (6) | 4 (4)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 6 (6) | 1 (1) | 3 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 2 (3) | 3 (3) | 3 (3) | 4 (4)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (5)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 5 (6) | 4 (4) | 5 (5) | 3 (3) | 4 (5)
NAUSEA (Gastrointestinal disorders) | 6 (6) | 4 (4) | 4 (4) | 12 (13) | 3 (4) | 10 (11) | 12 (12) | 20 (23)
VOMITING (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 3 (3) | 4 (5) | 4 (6) | 3 (3) | 5 (7)
FATIGUE (General disorders) | 2 (2) | 3 (3) | 4 (4) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 5 (5)
BACTERIAL VAGINOSIS (Infections and infestations) | 4 (4) | 4 (6) | 4 (5) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 4 (4) | 3 (3) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 4 (5)
SINUSITIS (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 5 (5) | 2 (2) | 2 (2) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (2) | 3 (3) | 1 (1) | 1 (2) | 0 (0) | 4 (6) | 2 (2) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (3) | 5 (7) | 4 (4) | 5 (5) | 1 (1) | 2 (2) | 2 (2)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
BLOOD CHOLESTEROL INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (5) | 2 (2)
BONE DENSITY DECREASED (Investigations) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
LIPIDS INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (6) | 3 (3) | 0 (0) | 3 (3) | 5 (5) | 4 (4) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5) | 2 (2) | 3 (3) | 2 (2) | 6 (7) | 6 (7) | 7 (7)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (4) | 5 (5) | 1 (1) | 3 (3)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
DIZZINESS (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1) | 3 (3) | 3 (4) | 3 (3) | 4 (5) | 5 (5)
HEADACHE (Nervous system disorders) | 6 (7) | 8 (8) | 9 (9) | 13 (14) | 8 (9) | 13 (15) | 11 (11) | 14 (14)
INSOMNIA (Psychiatric disorders) | 1 (1) | 7 (7) | 5 (5) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 5 (5)
DYSMENORRHOEA (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 5 (6) | 3 (4)
MENORRHAGIA (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 3 (3) | 4 (6) | 2 (2) | 1 (1) | 2 (2) | 7 (8)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
HOT FLUSH (Vascular disorders) | 2 (2) | 29 (32) | 16 (16) | 7 (7) | 4 (4) | 38 (39) | 14 (14) | 11 (11)
HYPERTENSION (Vascular disorders) | 3 (3) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 5 (6) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.